CLINICAL TRIAL: NCT00751257
Title: A Randomized Controlled Trial of Oral N-acetylcysteine for Smoking Reduction: a Pilot Study
Brief Title: N-Acetylcysteine and Smoking Reduction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Steven D. LaRowe, Ph.D.; Research Assistant Professor, Principal Investigator, Medical Univeristy of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P50DA015369 (NIH); P50DA015369 (NIH)
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2008-09

CONDITIONS: Nicotine Dependence
Keywords: Nicotine; N-acetylcysteine; smoking reduction
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Reduction | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 2400mg N-acetylcysteine (1200mg b.i.d.) for 4 consecutive weeks
  Interventions: Drug: N-acetylcysteine
- 2 (Placebo Comparator): Identically appearing placebo pills, packaged in an N-acetylcysteine "slurry" so that placebo will retain smell similar to active NAC capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — 2400mg (1200mg b.i.d., 600mg capsules, p.o.)
  Arms: 1
Drug: Placebo — Identically appearing placebo capsules, packaged in an N-acetylcysteine "slurry" so that placebo has similar odor as active NAC capsules
  Arms: 2

SUMMARY:
N-acetylcysteine is an inexpensive agent with a benign side effect profile with preliminary studies in humans suggesting efficacy for the treatment of cocaine dependence. N-acetylcysteine has been used in clinical medicine for nearly three decades to treat chronic lung conditions, acetaminophen overdose, and experimentally to treat cocaine dependence. It is generally safe and well tolerated. The present pilot study seeks to explore safety and tolerability, ad lib smoking, visual cue reactivity, and smoking reduction rates in a group of nontreatment seeking, nicotine dependence smokers who are willing to undergo a brief trial with oral N-acetylcysteine 1200 mg twice daily.

ELIGIBILITY:
Inclusion Criteria:

1. Be smokers motivated to reduce their cigarette usage but not seeking treatment to quit smoking at the time of screening.
2. Be Able to give written informed consent after being presented with an IRB-approved informed consent document
3. Be male or female of any race, between eighteen and sixty five years of age.
4. Be in stable physical and mental health as judged by interview
5. Be smoking 10 or more cigarettes per day for one or more years
6. Have an expired CO reading of ≥10 parts/million prior to beginning study
7. Test non-pregnant and use adequate birth control (female only). All female subjects will have a urine pregnancy test performed prior to the first dose of study medication.
8. Be able to comply with protocol requirements and be likely to complete all study treatments.
9. Live within 50 miles of the study site

Exclusion Criteria:

1. Have current dependence, defined by DSM IV criteria, on any psychoactive substance other than nicotine, alcohol, or marijuana or physiological dependence on alcohol requiring medical detoxification.
2. Have a history of significant hepatic, renal, endocrine, cardiac (i.e., arrhythmia requiring medication, angina pectoris, myocardial infarction,), stroke, seizure, neurological, non-drug-related psychiatric, gastrointestinal, pulmonary, hematologic or metabolic disorders.
3. Have a history of adverse reaction/hypersensitivity to N-acetylcysteine.
4. Have any significant active medical or psychiatric illness (e.g. schizophrenia, suicidal/homicidal ideation within the past 30 days) which might inhibit their ability to complete the study or might be complicated by administration of NAC.
5. Used carbamazepine or Nitroglycerin within the last 14 days or any other medication felt to be hazardous if taken with NAC
6. Have a current or past history of asthma and/or the occasional or daily use of Albuterol or other beta-agonist inhalers.
7. Females pregnant or breast-feeding
8. Have any medical history or condition considered by the investigator(s) to place the subjects at increased risk.
9. Not fail to actively meet the inclusion criteria at the time of screening.
10. Have a history of childhood or adult seizures of any cause.
11. Be currently taking any medications (i.e., beta-blockers, stimulant medications) that might affect heart rate or skin conductance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Carbon Monoxide Levels | Weekly
Smoking Level | Weekly
Craving Levels (Questionnaire for Smoking Urges -- Brief) | Weekly
Minnesota Nicotine Withdrawal Scale (MNWS) | Weekly

SECONDARY OUTCOMES:
Smoking Level | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Steven LaRowe, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States